CLINICAL TRIAL: NCT03558217
Title: Comparing Direct Anterior and Lateral Surgical Approaches for Collared and Collarless Implants and Correlating Joint Motion to Hip Implant Performance
Brief Title: Collared Versus Collarless Femoral Implants for Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Brent Lanting, Orthopaedic Surgeon, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 109401
Record Dates: First submitted 2017-11-17; First posted 2018-06-15 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2022-02

CONDITIONS: Hip Osteoarthritis; Hip Arthroplasty
Keywords: total hip arthroplasty; collarless femoral implant; collared femoral implant; direct anterior approach; direct lateral approach
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to have either the collared or collarless Corail femoral implant used during surgery and randomization will be stratified by surgical approach (determined by surgeon expertise).
Who Masked: Participant
Masking Description: Participants will be blinded to which group they have been assigned to until the final study visit at which point study personnel will reveal the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collared Femoral Implant (Experimental): Participants will have the Corail collared femoral implant used during their surgery.
  Interventions: Device: Collared Femoral Implant
- Collarless Femoral Implant (Active Comparator): Participants will have the Corail collarless femoral implant used during their surgery.
  Interventions: Device: Collarless Femoral Implant

INTERVENTIONS:
Device: Collared Femoral Implant — Corail collared femoral implant for total hip arthroplasty
  Arms: Collared Femoral Implant
Device: Collarless Femoral Implant — Corail collarless femoral implant for total hip arthroplasty
  Arms: Collarless Femoral Implant

SUMMARY:
This is a randomized control trial that will investigate whether a collared hip replacement implant provides greater stability compared to a collarless option. Stability will be measured by implant migration with radiostereometric analysis (RSA) imaging. Secondary objectives will be to compare function, quality of life and cost between the two implant types. We will also compare between two different surgical approaches, the direct anterior and direct lateral.

DETAILED DESCRIPTION:
Total hip arthroplasty (THA) is a procedure that has been demonstrated to provide excellent patient satisfaction and improve quality of life while being cost effective. The number of THA's conducted worldwide is expected to continue to grow; in some projections to grow exponentially. However, the environment for health care continues to evolve. Patients continue to demand higher activity levels, decreased recovery times, and greater patient autonomy. Health care economics are increasingly influencing clinical decision making. Bundled health care payments and more stringent evaluations are becoming the norm. Changes in care pathways based on patient input as well as due to health care economics are our new reality.

These two pervasive forces of change have led to a variety of care challenges and thought leaders have proposed solutions to these challenges. One solution that has responded to both changing patient expectations in their THA experience as well as the economic pressures has been rapid recovery pathways. An increase in rapid recovery care pathways and the growing prevalence of outpatient surgery and surgi-centers has enabled patients to increase their autonomy as well as decrease their time away from activities that are important to them such as employment. Rapid recovery care pathways also provide substantial cost savings by diminishing or eliminating inpatient care as well as enabling improved bed management options.

To facilitate rapid recovery programs, a variety of surgical changes have been made. Improved peri-operative care, decreased muscle trauma, improved hemostasis, and multi-modal analgesia have all made positive impacts. The increasing adaptation of the Direct Anterior Approach (DAA) relative to the Direct Lateral Approach (DLA) can be seen as a response to the need for rapid recovery programs as DAA has been demonstrated to enable earlier function and is thought to result in better patient outcomes, less pain, and shorter recovery times. Orthopaedic industry partners have also supported this change in practice by providing improved instrumentation and technologies to potentiate this minimal invasive surgical approach. A key change is the increasing use of implants that facilitate muscle sparing approaches: femoral components that do no require straight femoral reamers as well as broaches and implants with design features such as an angled lateral shoulder, abbreviated stem lengths, easy to control stem tips, and stems that do not require aggressive impaction to create intimate cortical contact. The Corail both has these features that potentiate surgery as well as excellent survivorship on registry and prospective studies.

In addition to the design features that potentiate minimally invasive implantation, the Corail stem has two main designs - the collared and collarless versions. Without question, the collar provides improved axial stability, and it has also been shown to provide improved rotational stability. It is unclear if this stability enables improved early function by providing the patient the sense that their implant is more stable immediately after surgery. Clinicians also appreciate the ability to more precisely control leg length during THA by ensuring the appropriate leg length is maintained when the collar abuts the calcar. The collar is felt to enable greater initial stability to the hip and provide the surgeon with greater confidence that the patient can embark on a rapid recovery care pathway.

However, not all surgeons are as supportive of implants that have a collar nor are they supportive of implants that have a collar, and highlight a lack of literature that is able to demonstrate the benefits. A lack of literature makes it a challenge for surgeons to adopt the change in philosophy. The purpose of this study is to examine the role of surgical approach and implant design on activity and implant fixation following THA.

ELIGIBILITY:
Inclusion Criteria:

* unilateral hip osteoarthritis
* primary total hip arthroplasty

Exclusion Criteria:

* symptomatic osteoarthritis in the contralateral hip
* bilateral total hip arthroplasty
* revision arthroplasty
* cognitive defects/neuromuscular disorders
* inability to understand English (questionnaires are only provided in English)
* live more than 100km from London, Ontario
* BMI greater than 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Implant Migration | 2 years
  Movement of the implant measured by radiostereometric imaging analysis.

SECONDARY OUTCOMES:
Timed-Up-and-Go (TUG) Test | baseline and 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years
  Measure to assess function.
Activity Level | baseline and 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years
  Activity measured by number of steps taken per day with the use of a FitBit.
University of California, Los Angeles (UCLA) Activity Score | baseline and 2 weeks, 4 weeks, 6 weeks, 3 months, 6 months, 1 year and 2 years
  Patient-reported outcome to assess activity level.
12-Item Short Form Health Survey (SF-12) | baseline and 3 months, 6 months, 1 year and 2 years
  General health questionnaire. Patient-reported measure to assess quality of life. Scores are calculated based on population averages.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | baseline and 3 months, 6 months, 1 year and 2 years
  Used to assess impact of hip and knee osteoarthritis. Patient-reported measure to assess function, pain and stiffness. Higher scores indicate worse pain, stiffness and functional limitations. Scores are separated into 3 subscales: pain, stiffness and function; but can be combined for a total score.
Harris Hip Score | baseline and 3 months, 6 months, 1 year and 2 years.
  Used to assess impact of hip osteoarthritis. Clinician-reported outcome measure to assess function, pain and range of motion. Higher scores indicate better outcomes and hip function.
EuroQol-5D (EQ-5D) | baseline and 6 weeks, 3 months, 6 months and 1 year
  Used to assess health-related quality of life. Patient-reported measure to assess quality of life.
Cost Questionnaires | 6 weeks, 3 months, 6 months and 1 year
  Patient-reported measure to assess indirect and direct costs of treatment including ER visits, clinician visits, tests and procedures, lost productivity, caregiver involvement, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Brent A Lanting, MD, FRCSC, Principal Investigator — London Health Sciences Centre
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Polus JS, Vasarhelyi EM, Lanting BA, Teeter MG. Acetabular cup fixation with and without screws following primary total hip arthroplasty: migration evaluated by radiostereometric analysis. Hip Int. 2024 Jan;34(1):42-48. doi: 10.1177/11207000231164711. Epub 2023 Apr 5. PMID 37016808